CLINICAL TRIAL: NCT01530997
Title: Phase II Study of De-intensification of Radiation and Chemotherapy for Low-Risk HPV-related Oropharyngeal Squamous Cell Carcinoma
Brief Title: De-intensification of Radiation & Chemotherapy in Low-Risk Human Papillomavirus-related Oropharyngeal Squamous Cell Ca
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1120
Record Dates: First submitted 2012-01-20; First posted 2012-02-10 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms
Keywords: Human Papilloma Virus; Oropharynx; Oropharyngeal Squamous Cell Carcinoma; Squamous Cell Carcinoma; Radiation Therapy; Chemotherapy; p16
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- De-escalated Radiation and Chemotherapy (Experimental): Patients will receive 54 to 60 Gy of Intensity Modulated Radiotherapy (IMRT) with concurrent weekly intravenous cisplatin (30 mg/m2). Diagnostic imaging (CT and/or MRI) will be obtained 4 to 8 weeks after completion of CRT to assess response. All patients will have surgical resection of any clinically apparent residual primary tumor or biopsy of the primary site if there is no evidence of residual tumor and will undergo a limited neck dissection to encompass at least those nodal level(s) that were positive pre-treatment, 4 to 14 weeks after CRT.
  Interventions: Radiation: Intensity Modulated Radiotherapy (IMRT); Drug: Cisplatin; Procedure: Limited surgical evaluation

INTERVENTIONS:
Radiation: Intensity Modulated Radiotherapy (IMRT) — All patients will receive IMRT. Dose painting IMRT will be used and all doses will be specified to the planning target volume (PTV). The high risk planning target volume (PTV-HR) and standard risk planning target volume (PTV-SR) will be treated to the following respective total doses: 60 Gy and 54 Gy. The dose per fraction to the PTV-HR and PTV-SR will be 2 Gy per day and 1.8 Gy per day, respectively. The PTV-HR will include the gross tumor and the PTV-SR will include the lymph nodes at risk for harboring micro-metastatic disease (i.e. subclinical disease).
Drug: Cisplatin — Cisplatin, 30mg/m2, will be given intravenously over 60 minutes weekly during IMRT; 6 total doses for a total of 180 mg/m2. It is preferred that the doses be administered on days 1, 8, 15, 22, and 29, and 36 of IMRT; however, this is not mandatory.
  Other Names: Platinol
Procedure: Limited surgical evaluation — 4 to 14 weeks after completion of CRT, patients will have at least a biopsy of the primary tumor and limited neck surgery to remove those lymph nodes that were involved with cancer prior to CRT.

SUMMARY:
The purpose of this research study is to learn about the effectiveness of using lower-intensity radiation and chemotherapy to treat human papillomavirus (HPV) associated low-risk oropharyngeal and/or unknown primary squamous cell carcinomas of the head and neck. The cure rate for this type of cancer is estimated to be high, > 90%. The standard treatment for this cancer is 7 weeks of radiation with 3 high doses of cisplatin. Sometimes surgery is performed afterwards. This standard regimen causes a lot of side effects and long term complications. This study is evaluating whether a lower dose of radiation and chemotherapy may provide a similar cure rate as the longer, more intensive standard regimen. Patients in this study will receive 1 less week of radiation and a lower weekly dose of chemotherapy followed by a limited surgical evaluation.

DETAILED DESCRIPTION:
The aim is to evaluate the pathological response rate of HPV positive and/or p16 positive low-risk oropharyngeal squamous cell carcinoma (OPSCC) after de-intensified chemoradiotherapy (CRT). Patients will receive 54 to 60 Gy of Intensity Modulated Radiotherapy (IMRT) with concurrent weekly intravenous cisplatin (30 mg/m2). Diagnostic imaging (CT and/or MRI) will be obtained 4 to 8 weeks after completion of CRT to assess response. All patients will have surgical resection of any clinically apparent residual primary tumor or biopsy of the primary site if there is no evidence of residual tumor and will undergo a limited neck dissection to encompass at least those nodal level(s) that were positive pre-treatment, 4 to 14 weeks after CRT. The primary endpoint of this study is the rate of pathological complete response (pCR) after CRT. Longitudinal assessments of quality of life and patient reported outcomes will be obtained prior to, during, and after CRT.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. T0-3, N0 to N2c, M0 squamous cell carcinoma of the oropharynx
3. Biopsy proven squamous cell carcinoma that is HPV and/or p16 positive
4. ≤ 10 pack-years smoking history or > 5 years of abstinence from smoking
5. History/physical examination within 8 weeks prior to registration
6. Radiologic confirmation of the absence of hematogenous metastasis within 12 weeks prior to registration.
7. The Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
8. Complete Blood Count (CBC)/differential obtained within 4 weeks prior to registration, with adequate bone marrow function defined as follows: Absolute neutrophil count (ANC) ≥ 1,800 cells/mm3; Platelets ≥ 100,000 cells/mm3; Hemoglobin ≥ 8.0 g/dl.
9. Adequate renal and hepatic function within 4 weeks prior to registration, defined as follows: Serum creatinine < 2.0 mg/dl; Total bilirubin < 2 x the institutional upper limit of normal (ULN); aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 3 x the institutional ULN.
10. Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential.
11. Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment.
12. Patients must be deemed able to comply with the treatment plan and follow-up schedule.
13. Patients must provide study specific informed consent prior to study entry.

Exclusion Criteria:

1. Prior history of radiation therapy to the head and neck
2. Prior history of head and neck cancer.
3. Severe, active co-morbidity, defined as follows: Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; Transmural myocardial infarction within the last 6 months; Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; Note, however, coagulation parameters are not required for entry into this protocol; Pre-existing ≥ grade 2 neuropathy; Prior organ transplant.
4. Known HIV positive
5. Significant pre-existing hearing loss, as defined by the patient or treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhishamjit Chera, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - Penrose Cancer Center, Colorado Springs, Colorado
  - University of Florida, Department of Radiation Oncology, Gainesville, Florida
  - University of North Carolina at Chapel Hill, Department of Radiation Oncology, Chapel Hill, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Rex Cancer Center of Wakefield, Raleigh, North Carolina

REFERENCES:
- [Background] Ang KK, Harris J, Wheeler R, Weber R, Rosenthal DI, Nguyen-Tan PF, Westra WH, Chung CH, Jordan RC, Lu C, Kim H, Axelrod R, Silverman CC, Redmond KP, Gillison ML. Human papillomavirus and survival of patients with oropharyngeal cancer. N Engl J Med. 2010 Jul 1;363(1):24-35. doi: 10.1056/NEJMoa0912217. Epub 2010 Jun 7. PMID 20530316
- [Derived] Mavroidis P, Price A, Fried D, Kostich M, Amdur R, Mendenhall W, Liu C, Das S, Marks LB, Chera B. Dose-volume toxicity modeling for de-intensified chemo-radiation therapy for HPV-positive oropharynx cancer. Radiother Oncol. 2017 Aug;124(2):240-247. doi: 10.1016/j.radonc.2017.06.020. Epub 2017 Jul 13. PMID 28712533
- [Derived] Chera BS, Amdur RJ, Tepper J, Qaqish B, Green R, Aumer SL, Hayes N, Weiss J, Grilley-Olson J, Zanation A, Hackman T, Funkhouser W, Sheets N, Weissler M, Mendenhall W. Phase 2 Trial of De-intensified Chemoradiation Therapy for Favorable-Risk Human Papillomavirus-Associated Oropharyngeal Squamous Cell Carcinoma. Int J Radiat Oncol Biol Phys. 2015 Dec 1;93(5):976-85. doi: 10.1016/j.ijrobp.2015.08.033. Epub 2015 Aug 22. PMID 26581135
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT01530997?term=LCCC1120&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrolling institutions included University of North Carolina Hospitals (Chapel Hill, NC), University of Florida Hospitals (Gainesville, FL), and Rex Hospital (Raleigh, NC).
Pre-assignment Details: Sixty-nine patients were eligible for enrollment, of whom 45 were accrued. One patient had a cerebrovascular accident during de-intensified CRT and was taken off the study. After the completion of CRT, 1 patient refused the planned surgical evaluation, leaving 43 patients who were fully evaluable.
Groups:
- Single Intervention: Patients received 60 Gy of Intensity Modulated Radiotherapy (IMRT) with concurrent weekly intravenous cisplatin (30 mg/m2). Diagnostic imaging (CT and/or MRI) was obtained 4 to 8 weeks after completion of CRT to assess response. Patients received surgical resection of any clinically apparent residual primary tumor or biopsy of the primary site if there was no evidence of residual tumor and underwent a limited neck dissection to encompass at least those nodal level(s) that were positive pre-treatment, 4 to 14 weeks after CRT.
  Intensity Modulated Radiotherapy (IMRT): All patients received IMRT. Dose painting IMRT was used and all doses were specified to the planning target volume (PTV). The high risk planning target volume (PTV-HR) and standard risk planning target volume (PTV-SR) was treated to the following respective total doses: 60 Gy and 54 Gy. The dose per fraction to the PTV-HR and PTV-SR was 2 Gy/day and 1.8 Gy/day, respectively.
Period: Overall Study
Arm/Group | Single Intervention
Started | 45
Completed | 43
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Sixty-nine patients were eligible for enrollment, of whom 45 were accrued. One patient had a cerebrovascular accident during de-intensified CRT and was taken off the study leaving 44 patients included in the baseline characteristics.
Groups:
- De-escalated Radiation and Chemotherapy: Patients received 60 Gy of Intensity Modulated Radiotherapy (IMRT) with concurrent weekly intravenous cisplatin (30 mg/m2). Diagnostic imaging (CT and/or MRI) was obtained 4 to 8 weeks after completion of CRT to assess response. Patients received surgical resection of any clinically apparent residual primary tumor or biopsy of the primary site if there was no evidence of residual tumor and underwent a limited neck dissection to encompass at least those nodal level(s) that were positive pre-treatment, 4 to 14 weeks after CRT.
  Intensity Modulated Radiotherapy (IMRT): All patients received IMRT. Dose painting IMRT was used and all doses were specified to the planning target volume (PTV). The high risk planning target volume (PTV-HR) and standard risk planning target volume (PTV-SR) was treated to the following respective total doses: 60 Gy and 54 Gy. The dose per fraction to the PTV-HR and PTV-SR was 2 Gy/day and 1.8 Gy/day, respectively.
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 44
Age, Continuous [Mean (Full Range); unit: years] | 61 [44 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 44
Marital Status [Count of Participants; unit: Participants]
  Married | 34
  Unmarried | 10
Tobacco Use [Count of Participants; unit: Participants]
  Never Smoker | 36
  <=10 Pack Years | 6
  > 10 Pack Years | 2
Primary Tumor Location [Count of Participants; unit: Participants]
  Tonsil | 16
  Base of Tongue | 26
  Unknown Primary | 2
T Stage [Count of Participants; unit: Participants] — The Classification of Malignant Tumours (TNM) system is the most widely used cancer staging system. The T refers to the size and extent of the main tumor. N refers to the regional lymph nodes. N0 means there is no cancer in nearby lymph nodes. The larger the number following N means the more lymph nodes that contain cancer.
  Participants
    T0 | 2
    T1 | 13
    T2 | 22
    T3 | 7
N Stage [Count of Participants; unit: Participants] — The Classification of Malignant Tumours (TNM) system is the most widely used cancer staging system. The T refers to the size and extent of the main tumor. N refers to the regional lymph nodes. N0 means there is no cancer in nearby lymph nodes. The larger the number following N means the more lymph nodes that contain cancer.
  Participants
    N0 | 4
    N1 | 10
    N2a | 2
    N2b | 21
    N2c | 7
HPV/p16 Status [Count of Participants; unit: Participants] — Human papilloma virus (HPV) is a common virus that can cause cancer. p16 is a tumor suppression gene that acts as a cyclin-dependent kinase inhibitor. HPV-related cancers with p16 overexpression (p16+) have a better prognosis than those not related to HPV due to an increased sensitivity to radiotherapy.
  Participants
    HPV+/p16+ | 28
    HPV-/p16+ | 16

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate After De-escalated CRT in HPV-positive and/or p16 Positive Oropharyngeal Squamous Cell Carcinoma (OPSCC).
Description: Pathologic Complete Response Rate is defined as no evidence of residual viable cancer in the evaluated pathological specimens.
Time Frame: 6 to 14 weeks after the last patient is enrolled, or approximately 24 to 32 months after study being opened
Population: Following the completion of chemoradiation therapy (CRT), 1 patient refused the planned surgical evaluation and 43 patients were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 43
Participants | 37

2. Secondary Outcome: Two-Year Local Control
Description: Local control is the arrest of cancer growth at the site of origin.
Time Frame: Median follow-up was 36 months with a range of 5-53 months
Measure: Number; unit: percentage of participants
Arm/Group | De-escalated Radiation and Chemotherapy
Number analyzed (Participants) | 44
percentage of participants | 100

3. Secondary Outcome: Regional Control
Description: Regional control is the percentage of participants who displayed control of cancer in sites that represent the first stages of spread from the local origin.
Time Frame: Median follow-up was 36 months with a range of 5-53 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Intervention
Number analyzed (Participants) | 44
percentage of participants | 100

4. Secondary Outcome: Cause-Specific Survival
Description: Cause-specific survival is the percentage of participants who have not died from low-risk low-risk OPSCC.
Time Frame: The median follow-up was 36 months with a range of 5-53 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Intervention
Number analyzed (Participants) | 44
percentage of participants | 100

5. Secondary Outcome: Distant Metastases Free Survival
Description: Distant metastases free survival is the percentage of subjects in a study who have survived without cancer spread.
Time Frame: the median follow-up was 36 months with a range of
Measure: Number; unit: percentage of participants
Arm/Group | Single Intervention
Number analyzed (Participants) | 44
percentage of participants | 100

6. Secondary Outcome: Overall Survival Rate
Description: The percentage of participants who are still alive from the start of treatment.
Time Frame: Median follow-up was 36 months with a range of 5-53 months.
Measure: Number; unit: percentage of participants
Arm/Group | Single Intervention
Number analyzed (Participants) | 44
percentage of participants | 95

7. Secondary Outcome: European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-H&N-35
Description: The head & neck cancer module of the EORTC QLQ comprises 35 questions assessing symptoms and side effects of treatment, social function and body image/sexuality.
  The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); several single item questions (Pain killers, nutritional supplements, feeding tube, weight loss, and weight gain) were just coded as no=1, yes=2. The scores of these scales were averaged from the scores of the component items, transformed and analyzed on a 0 - 100 scale. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning).
Time Frame: Prior to CRT, 4-8 weeks after CRT, follow-up visits for 2 years after CRT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Baseline: This data was collected pre-chemoradiotherapy treatment.
- 6-8 Weeks Post-Treatment: This data was collected 6-8 weeks post-chemoradiotherapy.
- Post-Surgery: This data was collected at the first follow-up post-surgery.
Arm/Group | Baseline | 6-8 Weeks Post-Treatment | Post-Surgery
Number analyzed (Participants) | 44 | 42 | 42
units on a scale
  Pain | 19 [14 to 25] | 25 [18 to 32] | 26 [20 to 33]
  Swallowing | 11 [7 to 14] | 19 [13 to 25] | 18 [13 to 24]
  Senses Problems | 5 [2 to 8] | 35 [29 to 40] | 28 [22 to 34]
  Speech Problems | 10 [5 to 15] | 13 [8 to 18] | 16 [11 to 22]
  Trouble with Social Eating | 8 [5 to 11] | 29 [22 to 37] | 24 [18 to 31]
  Trouble with Social Contact | 5 [2 to 8] | 15 [9 to 20] | 8 [4 to 12]
  Less Sexuality | 13 [7 to 19] | 34 [24 to 45] | 23 [15 to 31]
  Teeth | 3 [0 to 6] | 10 [5 to 16] | 12 [6 to 18]
  Opening Mouth | 5 [1 to 8] | 15 [9 to 21] | 18 [12 to 25]
  Dry Mouth | 16 [10 to 22] | 69 [61 to 77] | 64 [56 to 72]
  Sticky Saliva | 6 [2 to 10] | 61 [51 to 72] | 49 [41 to 58]
  Cough | 17 [11 to 24] | 25 [17 to 34] | 22 [15 to 29]
  Felt Ill | 8 [3 to 12] | 20 [11 to 28] | 11 [5 to 17]
  Pain Killers | 34 [20 to 48] | 43 [28 to 58] | 33 [19 to 48]
  Nutritional Supplements | 39 [24 to 53] | 55 [40 to 70] | 40 [25 to 56]
  Feeding Tube | 0 [0 to 0] | 40 [25 to 56] | 17 [5 to 28]
  Weight Loss | 20 [8 to 33] | 38 [23 to 53] | 36 [21 to 50]
  Weight Gain | 25 [12 to 38] | 40 [25 to 56] | 10 [1 to 19]

8. Secondary Outcome: European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 Global Health Status/QoL
Description: The EORTC QLQ-C30 is a cancer-specific instrument with 30 questions which incorporates 9 multi-item scales: 5 functional scales (physical, role, cognitive, emotional, and social); 9 symptom scales (fatigue, pain, nausea and vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties); and a global health and quality-of-life scale. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). The scores of these scales were averaged from the scores of the component items, transformed and analyzed on a 0 - 100 scale. A higher score=better level of functioning or greater degree of symptoms.
Time Frame: Prior to CRT, 4-8 weeks after CRT, follow-up visits for 2 years after CRT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Baseline | 6-8 Weeks Post-Treatment | Post-Surgery
Number analyzed (Participants) | 44 | 42 | 42
units on a scale
  Global health status/QoL | 80 [75 to 85] | 61 [55 to 68] | 69 [64 to 75]
  Physical functioning | 96 [93 to 98] | 78 [72 to 84] | 85 [79 to 90]
  Role functioning | 96 [93 to 98] | 65 [57 to 74] | 77 [69 to 84]
  Emotional functioning | 77 [70 to 84] | 77 [70 to 84] | 84 [78 to 90]
  Cognitive functioning | 91 [87 to 95] | 86 [81 to 92] | 87 [82 to 92]
  Social functioning | 88 [83 to 93] | 66 [58 to 74] | 81 [75 to 87]
  Fatigue | 20 [14 to 25] | 42 [34 to 50] | 31 [26 to 37]
  Nausea and vomiting | 2 [0 to 3] | 13 [8 to 17] | 4 [1 to 6]
  Pain | 15 [10 to 21] | 21 [13 to 29] | 20 [13 to 27]
  Dyspnea | 5 [1 to 8] | 11 [5 to 17] | 6 [1 to 10]
  Insomnia | 23 [16 to 30] | 34 [25 to 43] | 23 [15 to 31]
  Appetite loss | 14 [8 to 19] | 40 [30 to 49] | 33 [24 to 42]
  Constipation | 12 [5 to 18] | 17 [10 to 23] | 16 [9 to 23]
  Diarrhea | 5 [1 to 8] | 4 [1 to 7] | 6 [2 to 10]
  Financial difficulties | 16 [8 to 24] | 28 [17 to 39] | 22 [14 to 30]

9. Secondary Outcome: The Eating Assessment Tool (EAT-10) Composite Score
Description: The EAT-10 is a 10 item, validated self-administered instrument for documenting dysphagia severity. This questionnaire uses symptom-specific scores to assess dysphasia with solids, liquids, and pills as well as the impact of dysphagia on mental, social, and physical health. Higher raw scores represent worse QoL. All items have a 0-4 scale where 0 represents no problem and 4 represents severe problem. Total score can range from 0 to 40.
Time Frame: Prior to CRT, 4-8 weeks after CRT, follow-up visits for 2 years after CRT
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Post-Surgery: This data was collected at the first follow-up post surgery.
Arm/Group | Baseline | 6-8 Weeks Post-Treatment | Post-Surgery
Number analyzed (Participants) | 43 | 41 | 42
units on a scale | 4 [2 to 5] | 13 [9 to 16] | 11 [8 to 14]

10. Secondary Outcome: The Rosenbek Penetration Aspiration Scale
Description: The Rosenbek Penetration Aspiration Scale will be used to quantify dysphagia. It is an 8-point, equal-appearing interval scale to describe penetration and aspiration events. The measure was used for thin substances, pureed substances, and solid substances.
  1. Material does not enter airway 2. Material enters the airway, remains above the vocal folds, and is ejected from the airway. 3. Material enters the airway, remains above the vocal folds, and is not ejected from the airway. 4. Material enters the airway, contacts the vocal folds, and is ejected from the airway. 5. Material enters the airway, contacts the vocal folds, and is not ejected from the airway. 6.Material enters the airway, passes below the vocal folds, and is ejected into the larynx or out of the airway. 7. Material enters the airway, passes below the vocal folds, and is not ejected from the trachea despite effort. 8. Material enters the airway, passes below the vocal folds, and no effort is made to eject.
Time Frame: Prior to CRT and 4-8 weeks after completion of CRT
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-treatment: This data was collected before the treatment.
- Post-treatment: This data was collected 4-8 weeks after chemoradiation therapy
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 37 | 31
units on a scale
  Thin Substances | 1.30 (.62) | 1.90 (1.83)
  Pureed Substances | 1.03 (0.16) | 1.19 (0.54)
  Solid Substances | 1.03 (0.16) | 1.03 (0.19)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Single Intervention
All-Cause Mortality (participants affected / at risk) | 1/45
Serious Adverse Events (participants affected / at risk) | 15/45
Other Adverse Events (participants affected / at risk) | 40/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Intervention (N=45)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Sepsis (Infections and infestations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — Pulmonary embolus/Blood clot
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — Bleeding
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Hematoma (Vascular disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Soft tissue infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 2
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Intervention (N=45)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 3
Alanine aminotransferase increased (Investigations) | 1
Allergic reaction (Immune system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 29
Anemia (Blood and lymphatic system disorders) | 3
Anorexia (Metabolism and nutrition disorders) | 31
Anxiety (Psychiatric disorders) | 19
Constipation (Gastrointestinal disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 5
Depression (Psychiatric disorders) | 14
Dermatitis radiation (Injury, poisoning and procedural complications) | 32
Dry mouth (Gastrointestinal disorders) | 32
Dysgeusia (Nervous system disorders) | 32
Dysphagia (Gastrointestinal disorders) | 32
Esophageal pain (Gastrointestinal disorders) | 1
Esophageal stenosis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 32
Fever (General disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Infusion site extravasation (General disorders) | 1
Middle ear inflammation (Ear and labyrinth disorders) | 1
Mucosal infection (Infections and infestations) | 1
Mucositis oral (Gastrointestinal disorders) | 34
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 28
Neck edema (General disorders) | 29
Neutrophil count decreased (Investigations) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2
Pain (General disorders) | 34
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 31
Platelet count decreased (Investigations) | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Salivary gland infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 2
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 4
Syncope (Nervous system disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 16
Trismus (Musculoskeletal and connective tissue disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Vagus nerve disorder (Nervous system disorders) | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 18
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 1
Lymphopenia (Investigations) | 1
Diarrea (Gastrointestinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Severely altered eating/swallowing
Infections and infestations - Other, specify (Infections and infestations) | 1 — Respiratory Infection

LIMITATIONS AND CAVEATS:
Per the protocol, affiliate sites will only report grade 3/4 and all fatal (grade 5) toxicities. 1/2 toxicities were not reported for affiliate sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days